CLINICAL TRIAL: NCT05290714
Title: The Effectiveness and Change Mechanisms of Mentalization Based Therapy for Children (MBT-C)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Bilgi University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other); Anna Freud National Centre for Children and Families (Other)
Responsible Party: Principal Investigator, Sibel Halfon, Associate Professor, Istanbul Bilgi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MBT-C Trial
Record Dates: First submitted 2022-02-26; First posted 2022-03-22 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Mental Disorder, Child
Keywords: mentalization; internalizing problems; externalizing problems; comorbid internalizing/externalizing problems
MeSH Terms: conditions — Neurodevelopmental Disorders | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mentalization Based Treatment for Children (MBT-C) (Experimental): Mentalization Based Therapy for Children (MBT-C) is a transdiagnostic time-limited (12 weekly sessions) and manualized treatment for children aged between 5 to 12 years old with the main aim of increasing mentalization and restoring epistemic trust. Parallel parental work takes place to increase parental mentalization.
  Interventions: Behavioral: Mentalization-Based Treatment for Children (MBT-C)
- Parenting and Social Skills Group (Active Comparator): Parenting groups will run for 12 weeks with 10 parents per group. They will involve activities to help parents develop effective parenting skills via working on a family genogram, providing information on child development, developing acceptance and empathy, setting boundaries and anger regulation.
  The social skills groups will run for 12 weeks and will be conducted with 10 children per group. They will involve activities on self-presentation, peer communication, play skills, empathy and anger management.
  Interventions: Behavioral: Parenting and Social Skills Group

INTERVENTIONS:
Behavioral: Mentalization-Based Treatment for Children (MBT-C) — MBT-C will involve 12 paralel individual sessions with the parents and children separately conducted by two different therapists.
  Arms: Mentalization Based Treatment for Children (MBT-C)
Behavioral: Parenting and Social Skills Group — Parenting/social skills groups will be co-led by two therapists and involve 12 group therapy sessions with the parents and their children separately (10 parents and children per group).
  Arms: Parenting and Social Skills Group

SUMMARY:
The main aim of the project is to investigate the effectiveness and change mechanisms of Mentalization Based Therapy for Children (MBT-C; Midgley et al., 2017). MBT-C is a transdiagnostic treatment for children aged between 5 to 12 years old with the main aim of increasing mentalization and restoring epistemic trust. Parallel parental work takes place to increase parental mentalization. This project will test the effectiveness of MBT-C in a parallel group single blind pragmatic Randomized Controlled Trial (pRCT) conducted in Turkey in comparison to a parenting and social skills group. The sample will include 240 children between 5-12 years old with internalizing and externalizing and comorbid internalizing/externalizing problems and their parents. During the study, the patients will be randomized to two arms, and the treatment's effectiveness will be investigated both at short (8th and 12th weeks) and long terms (24th and 36th week) to also assess relapse prevention. Thelarge sample size and the longitudinal evaluation of primary (decrease in problems), and secondary outcomes will enable the investigation of mediators and moderators.

This project will also undertake a rigorous psychotherapy process study within the RCT, examining for the first time, for which children and under what circumstances MBT-C may be most effective, meaningfully linking process with outcome. For this purpose, patients' baseline characteristics, especially attachment security and mentalization deficits that may interact with treatment outcome (moderators) and different dimensions of mentalization that develop over the course of the treatment (change mechanisms/mediators) will be assessed.

ELIGIBILITY:
Inclusion criteria

1. Child age 5 to 12 years old
2. Clinical levels of child internalizing, externalizing and comorbid internalizing/externalizing problems (clinical levels on CBCL)

Exclusion criteria Children

1. a clinical diagnosis of autistic spectrum disorders (ASD) (meets KSADS-PL threshold criteria)
2. severe intellectual impairment (below 5th percentile on KBIT-2)
3. a clinical diagnosis of psychosis (meets KSADS-PL threshold criteria)
4. severe conduct disorder (clinical range on CBCL DSM-Oriented Conduct Problems scale)
5. severe substance abuse and dependence (meets KSADS-PL threshold criteria)
6. acute risk of harm to self and others (KSADS-PL risk item scores = 3)
7. an emergency/crisis referral, where an immediate response to a significant risk is required

Parents

1. risk of psychotism (clinical on BSI psychotism scale)
2. severe intellectual impairment (below 5th percentile on KBIT-2)
3. severe substance abuse and dependence (positive case on BAPIRIT)
4. acute risk of harm to self and others (BSI item 9, 39 & 40 = 4)
5. an emergency/crisis referral, where an immediate response to a significant risk is required

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to 36th week on the Child Behavior Checklist (CBCL) | Baseline (T0), 8th week (T1), 12th week (T2), 24th week (T3), 36th week (T4)
  The Child Behavior Checklist (CBCL; Achenbach, 1991) is a widely used method of identifying problematic behaviors in children with two separate versions for ages 1.5-5 and 6-18. The CBCL asks the parents to indicate how true a series of 112 problem behavior items are for their child in the past two months on a 3-point likert scale (0 = "not true", 1= "sometimes true", and 2 = "very true or often true"). Outcomes can be determined for significant problems for Internalizing (e.g., depression, anxiety), Externalizing (e.g., aggression, violence) or Total Problems. The scale has been adapted to Turkish with good reliability and validity (Erol et al., 1995).

SECONDARY OUTCOMES:
Change from Baseline to 36th week on the Me and My Feelings Questionnaire (M&MF) | Baseline (T0), 8th week (T1), 12th week (T2), 24th week (T3), 36th week (T4)
  Me and My Feelings Questionnaire (M&MF; Deighton et al., 2013) is a child-report measure consisting of total short 16-items: 10-items of emotional difficulties scale and 6-items of behavioral difficulties scale. It is scored on a 3-point likert scale (0 = "never expressed", 1 = "sometimes expressed", 2 = "always expressed"). Total score of scales are calculated as the sum of item scores with threshold values 10 for the emotional difficulties and six for the behavioral difficulties. Higher scores of each set of difficulties indicate the probability of mental health problems. The scale has been adapted to Turkish with good reliability and validity (İlnem, 2020).
Change from Baseline to 36th week on the Emotion Regulation Checklist (ERC) | Baseline (T0), 8th week (T1), 12th week (T2), 24th week (T3), 36th week (T4)
  Emotion Regulation Checklist (ERC; Shields & Cicchetti, 1997) is a parent-report measure of children's emotion regulation characteristics and involves 24-items rated on a 5-point likert scale (1 = "never" to 5 = "always"). It taps into two factors one of which is emotional lability and negativity defined as arousal, anger dysregulation, and mood changes; and the second is emotion regulation defined as socially appropriate emotional displays, empathy, and emotional selfawareness. The scale has been adapted to Turkish with good reliability and validity (Batum & Yagmurlu, 2007).
Change from Baseline to 12th week on the Children's Global Assessment Scale (CGAS) | Baseline (T0), 8th week (T1), 12th week (T2)
  The Children's Global Assessment Scale (CGAS; Schaffer et al., 1983) is a numeric scale (from 1 to 100) used by mental health clinicians to rate the global functioning of children under the age of 18 on a scale of 0 to 100. 90-81 range is scored when there is "good functioning in all areas; security in family, school, and with peers with only transient difficulties and everyday worries"; 50-41, when there is "moderate degree of interference in functioning in most social areas or severe impairment of functioning in one area"; and 20-11, when there is "need for considerable supervision to prevent hurting others or self or to maintain personal hygiene or gross impairment in all forms of communication". The scale has been adapted to Turkish with good reliability and validity (Gökler et al., 2004).
Change from Baseline to 36th week on the Parental Stress Index - Short Form (PSI-SF) | Baseline (T0), 8th week (T1), 12th week (T2), 24th week (T3), 36th week (T4)
  Parental Stress Index - Short Form (PSI-SF; Abidin, 1983) is a 36-item parent-report scale.The PSI-SF contains 36 items divided into three subscales, each composed of 12 items: "Parental distress"; "Parent-child dysfunctional interaction"; "Difficult child". Each item is rated on a 5-point likert scale from 1 = "strongly disagree" to 5 = strongly agree". The PSI-SF gives three subscores and a total distress score. The scale has been adapted to Turkish with good reliability and validity (Mert et al., 2008).
Change from Baseline to 36th week on the Parent Reflective Functioning Questionnaire (PRF-Q) | Baseline (T0), 8th week (T1), 12th week (T2), 24th week (T3), 36th week (T4)
  Parental Reflective Functioning Questionnaire (PRFQ; Luyten et al. 2017) includes 18 items divided into three subscales that measure PRF. A 7-point likert scale from 1 (strongly disagree) to 7 (strongly agree) is used to score each item. The PRFQ gives three subscales pertaining to "curiosity and interest in mental states", "prementalizing modes" and "certainty about mental states". The scale is in the process of being adapted to Turkish by our research group.
Change from Baseline to 36th week on the Difficulties in Emotion Regulation Scale (DERS) | Baseline (T0), 8th week (T1), 12th week (T2), 24th week (T3), 36th week (T4)
  Difficulties in Emotion Regulation Scale (DERS; Gratz & Roemer, 2004) is an instrument measuring emotion regulation problems in adults (to be used with parents in the current study). The scale comprises 36 items that are rated on a 5-point likert scale from 1 = "almost never" to 5 = "almost always", with higher scores indicating a difficulty of emotion regulation. The scale produces scores on the following subscales: (a) lack of awareness of emotional responses; (b) lack of clarity of emotional responses; (c) nonacceptance of emotional responses; (d) limited access to effective strategies; (e) difficulties in controlling impulsive behavior when experiencing negative affect; and (f) difficulties in engaging goal directed behavior when experiencing negative affect as well as a total disregulation score. The scale has been adapted to Turkish with good reliability and validity (Yiğit & Güzey-Yiğit, 2017).

OTHER OUTCOMES:
Screening: Brief Symptom Inventory (BSI) | Baseline (T0)
  Parents' initial psychopathology levels will be screened by the Brief Symptom Inventory (BSI; Derogatis, 1992). The BSI is an 53 item self-report scale and assesses three symptom scales, covering nine symptom dimensions: Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism; and three global indices of distress: Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. Items are rated on a 5-point likert scale from 1 = "never" to 5 = "a lot". The Turkish adaptation of the scale was conducted by Şahin and Durak (1994).
Screening: Schedule for Affective Disorders and Schizophrenia for School Aged Children (6-18 Years) (K-SADS-PL DSM-5) | Baseline (T0)
  Schedule for Affective Disorders and Schizophrenia for School Aged Children (6-18 Years) (K-SADS-PL DSM 5; Kaufman et al., 2016) is a semi-structured interview that probes child psychiatric disorders according to DSM-5 criteria. If a primary symptom is endorsed, further questions are asked to determine whether diagnostic criteria are met. In the study, specific components of the instrument will be selected to screen for psychosis, autistic spectrum disorders, substance abuse and dependence, acute risk of harm to self and others. It was adapted to Turkish by Ünal et al. (2019).
Screening: Kaufman Brief Intelligence Test-Second Edition (KBIT-2) | Baseline (T0)
  Kaufman Brief Intelligence Test-Second Edition (KBIT-2, Kaufman & Kaufman, 1990) will be used to screen for general intelligence in children and their parents. The Verbal Scale contains two kinds of items-Verbal Knowledge and Riddles-both of which assess crystallized ability.The Nonverbal Scale includes a Matrices subtest that assesses fluid thinking-the ability to solve new problems by perceiving relationships and completing analogies. The KBIT-2 provides Verbal and Nonverbal Scores, plus a composite IQ. The scale was adapted to Turkish with good reliability and validity (Savasan, 2006).
Screening: BAPIRT Alcohol and Drug Questionnaire | Baseline (T0)
  BAPIRT Alcohol and Drug Questionnaire (Ogel et al., 2017) is a risk-screening questionnaire appropriate for Turkish cultural characteristics in detection of alcohol- and drug-use level through utilization of Addiction Profile Index (API). BAPİRT-alcohol and BAPİRT-drug subscales each involve 6 questions rated on a 3 point likert scale (0 = "none", 1 = "often", 2= "very frequently"). The scale was constructed for use in the Turkish culture by Öğel et al. (2017).
Baseline Moderator: Adverse Childhood Experiences Scale (ACE) | Baseline (T0)
  In order to measure parents' and children's early trauma history, an adapted version of the Adverse Childhood Experiences (ACE) questionnaire (Dube et al., 2003; Murphy et al., 2007) will be used. ACE is a parent-report scale and assesses retrospectively forms of abuse, neglect, and household dysfunction (i.e., witnessing domestic violence, separation and mental illness in the family) both for the parent's and child's early history. Scores range from 0-10 on the ACE, with the latter representing full exposure at some point in the first 18 years of life, to all forms of household dysfunction and abuse detailed in the questionnaire. The scale has been adapted to Turkish by Gunduz et al. (2018).
Baseline Moderator: Attachment Doll Story Completion Task (ASCT) | Baseline (T0)
  An adapted version of the Attachment Doll Story Completion Task (ASCT; Bretherton et al., 1990) will be used to assess the quality and the security of attachment-related representations of children's relationships with their caregivers. ASCT was originally designed for three-year-olds and later adapted to school age children by Granot and Mayseless (2001). ASCT comprises of five storystems that aim to elicit stories from children on attachment-related day-to-day issues. A set of family figure dolls and related props are used to prime children and invite them to complete unfinished stories. Children are classified as secure, fairly secure or insecure based on their responses. The scale was adapted to Turkish by Uluç (2005).
Baseline Moderator: Kerns Security Scale (KSS) | Baseline (T0)
  The Kerns Security Scale (KSS; Kerns et al., 1996) will be used to assess children's baseline attachment security. KSS is a child-report scale and comprises of 15 items measuring (a) the extent to which children believe that their attachment figures are sensitive and available; (b) their tendency to trust attachment figures under stress; and (c) their level of willingness to communicate with attachment figures. Children complete the form separately from both their mother and fathers. The items are rated on a 4-point likert scale "Some kids . . . Other kids. . ." format with higher scores indicating a more secure attachment. The scale was adapted to Turkish by Sümer and Anafarta-Şendağ (2009).
Baseline Moderator: Experiences in Close Relationships Scale-II (ECR-II) | Baseline (T0)
  Experiences in Close Relationships Scale-II (ECR-II; Fraley et al., 2000) will be used to assess the attachment patterns of the parents at baseline. The ECR-II consists of a total of 36 items, 18 in the anxiety and 18 in the avoidance sub-dimensions. The items are answered on a 7-point likert scale (1= "Never Agree", 7= "Strongly Agree"). The scores for each attachment dimension are calculated by taking the average of the item total score. The increase in scores indicates an increase in the anxious or avoidant attachment patterns. The adaptation study of the ECR-II Turkish Form was conducted by Selcuk et al. (2005).
Baseline Moderator: The Child Attachment Interview (CAI; Target et al. 2003) | Baseline (T0)
  The Child Attachment Interview (CAI; Target et al. 2003) is a 19-question, semi-structured interview for 8- to 12-year-olds that assesses children's attachment representations of their current relationships with their primary caregivers. CAI coders rate videotapes and verbatim transcripts on 11 9-point scales (e.g., idealization of attachment figures, balance of positive/negative references to attachment figures).
Experience of Service Questionnaire (ESQ) | 12th week (T2)
  The Experience of Service Questionnaire (ESQ, Brown et al., 2014) consists of 12 items rated on a 3-point likert scale (1 = "not true"; 3 = "certainly true") and 3 free text sections looking at what the respondent liked about the service, what they felt needed improving, and any other comments.
Therapeutic Alliance Scale for Children-revised (TASCr-C, TASCr-T, TASCr-P) | 3rd week (T1) 8th week (T2) 12th week (T3)
  The Therapeutic Alliance Scale for Children-revised (TASC-r, Shirk et al., 2011) will be used as a measure of therapeutic alliance across treatment. The TASC is a 12-item, 4-point Likert-type scale completed by the children and parents and there is a parallel version for the therapist to complete. Each item is rated on a 4 point scale ranging from 1 = "not at all" to 4 = "very much". The scale will be administered to patients in the MBT-C arm.

CONTACTS AND LOCATIONS:
Overall Officials: SİBEL HALFON, PhD, Principal Investigator — Istanbul Bilgi University
Locations (1):
- Istanbul Bilgi University Psychological Counseling Center, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
After publication of the primary objective, published data might be provided to interested scientists on request for meta-analyses or secondary analyses of variables of interest in an anonymized way, with permission from the trial team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the end of the study

REFERENCES:
- [Background] Midgley, N., Ensink, K., Lindqvist, K., Malberg, N., & Muller, N. (2017). Mentalization-based treatment for children: A time-limited approach. American Psychological Association. https://doi.org/10.1037/0000028-000